CLINICAL TRIAL: NCT02904278
Title: Randomized, Controlled Trial of a Novel Mobile Device Application to Improve Adherence in Children Greater Than 11 Years of Age After Cardiac Transplantation (CTOTC-10)
Brief Title: Novel Mobile Device Application to Improve Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation in Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DAIT CTOTC-10
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Pediatric Heart Transplant Recipients; Pediatric Cardiac Transplantation; Pediatric Heart Transplantation
Keywords: Mobile Application Intervention; Teen Pocket PATH® [TPP]; Adherence; Medical Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teen Pocket PATH® Mobile Application (Experimental): Participants in this group will receive the mobile application for improving adherence to their post-transplant medications, along with standard post-transplant care, in accordance with the CTOTC-10 Cardiac Consortium Clinical Care Guidelines.
  The intervention will prompt, remind, and warn participants when medications are due, inform parents when medication management is completed, and engage parents when no action is undertaken. Additionally, the mobile app. will inform the investigators, by way of automated text messaging, of treatment adherence.
  Duration of participation: up to 12 months post heart transplantation.
  Interventions: Other: Teen Pocket PATH® Mobile Application
- Control Group: Standard of Care (Other): Participants in the control group will receive standard post-transplant care, in accordance with the CTOTC-10 Cardiac Consortium Clinical Care Guidelines.
  Duration of participation: up to 12 months post heart transplantation.
  Interventions: Other: Control Group: Standard of Care

INTERVENTIONS:
Other: Teen Pocket PATH® Mobile Application — Participants in the intervention group will receive the mobile application for improving adherence to their post-transplant medications. The intervention will prompt, remind, and warn participants when medications are due, inform parents when medication management is completed, and engage parents when no action is undertaken.
  Other Names: TPP mobile app; Mobile health application; Mobile app; cell phone app
  Arms: Teen Pocket PATH® Mobile Application
Other: Control Group: Standard of Care — Adolescents and parents/guardians assigned to the Standard Care Condition will receive standard clinical care per standard site procedures.
  Other Names: Post Heart Transplant Standard of Care
  Arms: Control Group: Standard of Care

SUMMARY:
The purpose of this study is to collect and compare information on how and when adolescent heart transplant recipients take their prescribed medication. The investigators want to find out if regular use of 'an app' on cell phones, called the Teen Pocket PATH® (TPP), can help adolescents take their medication according to their prescribed dosing schedule. This may then help reduce complications of transplant, such as rejection. The investigators also want to find out if how adolescent heart transplant recipients take their medications affects the development of antibodies in their blood. Antibodies are small proteins in the blood that may develop after heart transplantation, and which can sometimes damage a new heart.

DETAILED DESCRIPTION:
This is a multi-center, randomized, open label clinical trial of a novel mobile application. The intervention in this randomized controlled trial is the provision of a novel mobile health application (Teen Pocket PATH® [TPP]). Participants will include heart recipients 11-17 years of age transplanted at one of the listed study sites (refer to Contacts and Locations Section of this ClinicalTrials.gov record).

It is important that heart transplant recipients take their prescribed heart transplant medication. One of the challenges for adolescent (children ages 11 to 17) heart transplant recipients is being able to follow their medication dosing schedule consistently. The purpose of this study is to collect and compare information on how and when adolescent heart transplant recipients take their prescribed medications. The investigators want to find out if regular use of 'an app' on the participant's cell phone, called the Teen Pocket PATH® (TPP), can help adolescent heart transplant recipients take their medication according to their prescribed dosing schedule. This may then help reduce complications of transplant, such as rejection. The investigators also want to evaluate whether how one takes their medications affects the development of antibodies in their blood. Antibodies are small proteins in the blood that may develop after heart transplantation, and which can sometimes damage a recipient's new heart.

The TPP app provides reminders to the participant and their parent/guardian, includes a list of their medications, and maintains a log to help track medication taking. The parent(s) will receive a text message when their participating child enters into the TPP app that s/he has taken his/her medication. The parent(s) will also be notified via text if their participating adolescent child does not enter information into the TPP app regarding their medication adherence and related timing information. The information collected on the TTP app will be available to the study investigators.

Eligible participants will be randomly selected (randomized) to be in one of two groups: this means that each participant will have an equal but random chance of being assigned to:

* the Experimental Group - participants will receive standard of care and use the TPP app to monitor how they take their medication or
* the Control Group - participants will receive standard of care and will not not receive the TPP app.

Both groups will have the same number of scheduled research visits and will receive the usual treatment and medication provided by their doctor for their heart transplant. Research visits will coincide with your routine clinic visits.

The study will not change the care that participants receive prior to, during or after transplantation. The study will collect information about participants, their medication dosing schedule, and their medical condition and care. In addition, the investigators will collect some blood at certain times for research. This blood will be used to measure antibodies in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled (consented) prior to hospital discharge from heart transplantation or within one month after discharge, but not later than 3 months post-transplantation;
* English as primary language or fluent in English; and
* Informed consent and assent obtained.

Exclusion Criteria:

* Positive donor-specific cytotoxicity requiring different immunosuppressive regimen from standard care;
* Inability or unwillingness of a participant to give written informed consent or comply with study protocol;
* Re-transplant or multi-organ transplant recipient;
* Condition or characteristic which in the opinion of the investigator makes the participant unlikely to complete at least one year of follow-up; or
* Current participation in other research studies that would, or might, interfere with the scientific integrity or safety of current study (e.g. by interference with immunosuppression management guidelines and study end-points).

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Variability in Tacrolimus Levels by Group Assignment | 3 months ( to 12 Months Post-Transplantation
  Variability in tacrolimus levels (standard deviation of post discharge first year outpatient tacrolimus levels commencing at 3 months post-transplantation).

SECONDARY OUTCOMES:
Count of Rejection Events within the First Year Post-Transplant by Group Assignment | Within 12 Months Post-Transplantation
  Rejection events will include acute cellular, mixed, and clinical rejection.
Count of Participants that Develop Post-Transplant De Novo Donor Specific Donor-Specific Antibody (DSA) and Autoantibodies by Group Assignment | Within12 Months Post-Transplantation
  De novo human leukocyte antigen (HLA) donor-specific antibodies (DSA), and antibodies to the self-antigens cardiac myosin and vimentin.
Comparison of Engagement in Self-Care Measured by the Medication Adherence Measure (MAM) by Group Assignment | At Baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 12 Months (Visit 4) Post-Transplantation
  Engagement in self-care as measured by self-report using the Medication Adherence Measure (MAM).
Engagement in Self-Care Measured by TPP Activity | Baseline (Visit 1), 3-months (Visit 2), 6 months (Visit 3), and 12 months (Visit 4) Post-Transplantation
  Engagement in self-care during the first year after heart transplantation as measured by the mobile app, Teen Pocket PATH® (TPP).
Comparison of Self-Reported Medication Adherence by Group Assignment | Baseline (Visit 1), 3-months (Visit 2), 6 months (Visit 3), and 12 months (Visit 4) Post-Transplantation
  Self-reported medication adherence assessed using the medication module of the Medication Adherence Measure (MAM).
  The MAM will be applied at each clinic visit unless within 7 days of prior visit. Scores for all surveys will be averaged over the course of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Shellmer, Ph.D., Study Chair — Children's Hospital of Pittsburgh: Pediatric Transplantation; Steven A. Webber, MBChB, MRCP, Principal Investigator — Monroe Carell Jr. Children's Hospital at Vanderbilt: Pediatric Transplantation
Locations (8):
- United States (8):
  - Emory University School of Medicine: Pediatric Transplantation, Atlanta, Georgia
  - Boston Children's Hospital: Pediatric Transplantation, Boston, Massachusetts
  - St. Louis Children's Hospital: Pediatric Transplantation, St Louis, Missouri
  - Columbia University Medical Center: Pediatric Transplantation, New York, New York
  - Montefiore Medical Center: Pediatric Transplantation, New York, New York
  - Children's Hospital of Philadelphia: Pediatric Transplantation, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh: Pediatric Transplantation, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt: Pediatric Transplantation, Nashville, Tennessee

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- See also: The National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: The Clinical Trials in Organ Transplantation in Children (CTOT-C) — http://www.ctotc.org/